CLINICAL TRIAL: NCT07403097
Title: Study of Autologous CD19-Targeted Chimeric Antigen Receptor T (CAR- T) Therapy for Refractory Systemic Lupus Erythematosus
Brief Title: Study of CD19 CAR-T Therapy for Refractory SLE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC098
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: CD19; CAR-T
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTOC1 (Experimental): This trial was designed as an open, single-arm, single-center, dose-exploration trial.
  Interventions: Biological: PTOC1

INTERVENTIONS:
Biological: PTOC1 — Three dose groups (1.5×10^5/kg, 5×10^5/kg,1×10^6/kg) were set up, starting from the low dose group climbing to explore the safe and effective dose.

SUMMARY:
This is an investigator-initiated trial aimed at assessing the safety and efficacy of PTOC1 cells Injection in the treatment of refractory systemic lupus erythematosus.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a serious autoimmune disease that can lead to extensive damage in multiple organs and systems, ultimately resulting in disability and even death.

Currently, the primary treatment for SLE relies on glucocorticoids and immunosuppressants to alleviate symptoms. However, due to the absence of a curative treatment, patients typically need to remain on medication indefinitely. In recent years, biological agents such as belimumab and rituximab have been introduced for the treatment of SLE, but these treatments cannot completely eliminate autoimmune B cells in the bone marrow, leading to unsatisfactory overall outcomes. In addition, discontinuing these drugs can lead to disease relapse, and patients still face the challenges of lifelong medication and an incurable disease.

CAR-T therapy is an adoptive cell therapy that uses genetic modification technology to reprogram T cells and eliminate target cells expressing disease-related antigens through antigen-specific recognition. Clinical studies have demonstrated that CD19-targeted CAR-T cells hold significant therapeutic potential for SLE. Compared with traditional CAR-T cells, PTOC1 cells Injection, relying on an innovative CAR-T manufacturing system, can be produced in an extremely short period of time (with a preparation time of only 10 minutes).

The purpose of this study is to assess the safety and efficacy of PTOC1 cells Injection in the treatment of refractory SLE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 5 years, no gender limitation;
* Diagnosed with SLE according to the 2019 EULAR/ACR classification criteria, and still in moderate to severe disease activity despite ≥ 3 months of high dose glucocorticoids(prednisone≥1mg/kg/d or other equivalent amount of other steroid), combined with hydroxychloroquine, and at least 2 Immunosuppressants or biologics (including cyclophosphamide, mycophenolate mofetil, azathioprine, methotrexate, cyclosporin, tacrolimus, sirolimus, leflunomide, telitacicept, belimumab, and rituximab) or intolerant to standard treatments;
* SLEDAI-2K score ≥ 8 points;
* The functions of vital organs must meet the following requirements:

  1. cardiac function: left ventricular ejection fraction (LVEF) ≥ 50%, with no obvious abnormalities on electrocardiogram (ECG);
  2. renal function: eGFR ≥ 30 mL/min/1.73m2;
  3. hepatic function: AST and ALT ≤ 3.0×ULN, total bilirubin ≤ 2.0×ULN;
  4. pulmonary function: no severe pulmonary lesions; blood oxygen saturation ≥ 92% under non-oxygen supplementation conditions.
* Meet the criteria of leukapheresis or intravenous blood collection, and no contraindication for leukapheresis;
* Negative pregnancy test for female subjects of childbearing age, and agree to take effective contraceptive measures until one year after infusion;
* Participant or his/her guardians agree to participate in the clinical trial and sign the informed consent form indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study.

Exclusion Criteria:

* Central nervous system (CNS) diseases: presence of CNS lupus symptoms requiring intervention within 60 days, including epilepsy, confusion, cerebrovascular events, etc;
* Congenital heart disease or severe arrhythmia before screening: Including multifocal and frequent supraventricular tachycardia, ventricular tachycardia, etc.; or complicated with moderate to large pericardial effusion, severe myocarditis, etc.; or patients with unstable vital signs who require vasopressors to maintain blood pressure;
* Presence of active infections requiring systemic treatment or uncontrolled infections within 3 months prior to screening;
* Having received solid organ transplantation or hematopoietic stem cell transplantation within 3 months prior to screening; or having grade 2 or above acute graft-versus-host disease (GVHD) within 2 weeks prior to screening;
* Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood hepatitis B virus (HBV) DNA level exceeding the normal range; positive for hepatitis C virus (HCV) antibody with peripheral blood hepatitis C virus (HCV) RNA level exceeding the normal range; positive for human immunodeficiency virus (HIV) antibody; positive for treponema pallidum antibody;
* History of macrophage activation syndrome within 1 month prior to screening (except for those for whom the investigator has determined that safety risks are excluded after treatment);
* History of previous CAR-T therapy (except for those for whom the investigator has determined that safety risks are excluded after treatment);
* Presence of active pulmonary tuberculosis at the time of screening;
* Having received any vaccination within 4 weeks prior to screening;
* Positive result of blood pregnancy test;
* A confirmed diagnosis of malignant diseases such as tumors prior to screening;
* Participation in other clinical trials within 3 months prior to enrollment;
* Other circumstances that the investigator deems inappropriate for participation in this study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The safety of PTOC1 cell therapy in patients with refractory SLE [Safety] | 3 months
  Types, frequency and severity of adverse events.
The changes in SLEDAI-2K from baseline [efficacy] | 6 months
  Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) ranges from 0 to 105 points. The higher the score, the higher the disease activity.
The changes in PGA from baseline [efficacy] | 6 months
  Physician Global Assessment(PGA) is a continuous visual analogue scale with 0, 1, 2, and 3 scores. "0" indicates no disease activity and "3" indicates the most severe disease activity.
The changes in BILAG-2004 from baseline [efficacy] | 6 months
  British Isles Lupus Assessment Group Index 2004(BILAG-2004) consists of 8 systems, each of which is graded as A, B, C and D. "A" indicates that the condition is highly active and requires active treatment. "B" indicates that the condition is active and requires close monitoring or symptomatic treatment. "C" indicates a stable condition. "D" indicates that the system is uninvolved.
The number of patients with SRI-4 response [efficacy] | 3 months
  The definition of SRI-4 response: SLEDAI-2K ≥ 4 points improvement; PGA <0.3 points increase; BILAG 2004 with no new A grade score and no more than 1 new B grade score.
The number of patients with LLDAS [efficacy] | 6 months
  The definition of LLDAS: SLEDAI-2K ≤ 4 points and no disease activity in major organs (kidney, central nervous system, heart and lung), and no vasculitis or fever; no new disease activity symptoms compared with previous disease assessments; PGA ≤ 1; serological parameters not required; with the permitted use of low-dose glucocorticoids (prednisolone ≤ 7.5 mg/day), and/or stable immunosuppressives and biologics.
The number of patients with DORIS [efficacy] | 6 months
  The definition of DORIS: SLEDAI-2K = 0 points; PGA < 0.5 points; serological parameters not required; with the permitted use of antimalarials, low-dose glucocorticoids (prednisolone ≤ 5 mg/day), and/or stable immunosuppressives and biologics.

SECONDARY OUTCOMES:
Cmax of PTOC1 cells [PK parameter] | 3 months
  The peak concentration (Cmax) of amplified PTOC1 cells in peripheral blood after infusion can be measured.
Tmax of PTOC1 cells [PK parameter] | 3 months
  The time for amplified PTOC1 cells in peripheral blood to reach the maximum concentration (Tmax) can be measured.
AUC28d/90d of PTOC1 cells [PK parameter] | 3 months
  The area under the plasma concentration-time curve from 28 to 90 days after infusion (AUC28d/90d) can be measured.
The degree of B cell depletion [PD parameter] | 3 months
  The degree of CD19+ B cell depletion at different time points.
The concentration of IL-6 [PD parameter] | 3 months
  The serum concentration of CAR-T therapy-related cytokines such as IL-6 at different time points.
The concentration of CRP [PD parameter] | 3 months
  The serum concentration of CAR-T therapy-related cytokines such as CRP at different time points.
The concentration of ferritin [PD parameter] | 3 months
  The serum concentration of CAR-T therapy-related cytokines such as ferritin at different time points.
The proportion of major B-cell subtypes | 6 months
  The proportion of major B-cell subtypes at each visit time point after infusion.
The correlation between the proportion of major B-cell subtypes and the reduction of disease activity | 6 months
  The correlation between the proportion of major B-cell subtypes at each visit time point after infusion and the reduction of disease activity relative to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, China